CLINICAL TRIAL: NCT05434195
Title: Clinical Antenatal Randomised Study to CharactErise Key Roles of TetrahydroFOLate in HyperTensive Pregnancies (CAREFOL-HT)
Brief Title: Clinical Antenatal Randomised Study to CharactErise Key Roles of TetrahydroFOLate in HyperTensive Pregnancies
Acronym: CAREFOL-HT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); British Heart Foundation (Other); Merck & Cie (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 295830
Record Dates: First submitted 2022-05-05; First posted 2022-06-27 (Actual); Last update posted 2022-06-27 (Actual); Status verified 2022-05

CONDITIONS: Pre-Eclampsia; Pregnancy Induced Hypertension; Pregnancy Related
Keywords: 5-methyltetrahydrofolate; Tetrahydrobiopterin; Pre-Eclampsia; Antenatal study
MeSH Terms: conditions — Pre-Eclampsia; Hypertension, Pregnancy-Induced

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Normotensive (No Intervention): A sub-cohort of 32 normotensive women will be recruited to establish normal pregnancy values for the measures performed as well as validation of outcome measures.
- Preeclampsia - Placebo (Placebo Comparator): A sub-cohort of 32 preeclampsia women will be recruited taking the placebo.
  Interventions: Dietary Supplement: Arcofolin® Placebo
- Preeclampsia - low dosage (Active Comparator): A sub-cohort of 32 preeclampsia women will be recruited taking the placebo low dose of 5-MTHF.
  Interventions: Dietary Supplement: Arcofolin® 5-Methyltetrahydrofolate
- Preeclampsia - high dosage (Active Comparator): A sub-cohort of 32 preeclampsia women will be recruited taking the placebo high dose of 5-MTHF.
  Interventions: Dietary Supplement: Arcofolin® 5-Methyltetrahydrofolate

INTERVENTIONS:
Dietary Supplement: Arcofolin® 5-Methyltetrahydrofolate — 5-methyltetrahydrofolate (5-MTHF) is the biologically active form of reduced folate, which can increase BH4 availability. 5-MTHF is available as a nutritional vitamin (Merck & Cie) for human use including during pregnancy. Two out of three preeclamptic study groups will receive 5-MTHF - one at a low dose and the other at a high dose.
  Other Names: Arcofolin®
  Arms: Preeclampsia - high dosage; Preeclampsia - low dosage
Dietary Supplement: Arcofolin® Placebo — The placebo, this consists of the same excipients as 5-MTHF, microcrystalline cellulose and silica with no active ingredient.
  Arms: Preeclampsia - Placebo

SUMMARY:
Study background

High blood pressure during pregnancy is a worldwide health problem that can be dangerous to mothers and commonly causes premature birth and small babies. There is also growing evidence that mothers who suffer from high blood pressure in pregnancy, and their babies, have a higher risk of high blood pressure and cardiovascular disease later in life. Previous studies have revealed detrimental changes in the structure and function of the heart and blood vessels of mothers, and their babies, who experience this common complication. These changes may explain their increased risk of later disease. The investigators have also learned through previous studies that tetrahydrobiopterin (BH4), a molecule that has a role in blood vessel health, plays an important role in stabilising blood vessel function. Lower levels of BH4 are evident in both the placenta and the umbilical cord from mothers with high blood pressure. We, therefore, want to investigate how closely BH4 levels are related to clinical features of pre-eclampsia and whether altering levels of BH4, using a nutritional supplement, improves features of the disease such as blood vessel function. To do this, the investigators need to compare the levels of BH4 between mothers with pre-eclampsia, those taking the supplement and those without pre-eclampsia. The investigators also compare how the heart and blood vessels look and function in these groups using ultrasound methods, including echocardiography and fetal sonography.

Study objectives

CAREFOL-HT will assess how levels of BH4 differ in pregnant women with high blood pressure and if this is reflected in functional changes in the heart and blood vessels of these women. The investigators will also determine whether changing levels of BH4, using a tetrahydrofolate supplement (5-MTHF), changes blood vessel function.

DETAILED DESCRIPTION:
High blood pressure during pregnancy is a world-wide health problem that can be dangerous to mothers, and commonly causes premature birth and small babies. There is also growing evidence that mothers who suffer from high blood pressure in pregnancy and their babies both have a higher risk of high blood pressure and cardiovascular disease in later life. Previous studies have revealed detrimental changes in the structure and function of the heart and blood vessels of mothers and their babies who experience this common complication which may be important in understanding the subsequent increased risk of later disease. The investigators have also learned through previous work carried out by our research group that certain biological processes may be disturbed in women with high blood pressure in pregnancy. One of these processes involves a molecule called tetrahydrobiopterin (also known as BH4) which is required for the correct functioning of blood vessels. Supplementation with biologically-active forms of reduced folate are able to increase the levels of this molecule and can reverse the changes caused by high blood pressure in pregnant mice, and in cultured human endothelial cells. These particular folate supplements are safe and approved for use in pregnancy, but are not widely used as they are more specialised and currently less available than folic acid, the oxidized form of folate that is widely used for supplementation in pregnancy. However, folic acid does not have the same effects as the specific biologically-active form of reduced folate (tetrahydrofolate), because folic acid requires enzymatic conversion within the body in order to generate the biologically-active form of reduced folate. Whilst the use of folic acid appears to be sufficient in most cases to increase folate levels in the prevention of fetal abnormalities such as neural tube defects, the conversion of folic acid to its biologically-active reduced form may be itself deficient or detrimental in women with preeclampsia, and does not increase tetrahydrobiopterin levels. Indeed, folic acid treatment has been found to be ineffective in a large clinical trial to improve high blood pressure in pregnancy women.

This clinical trial will investigate the levels of biologically-active forms of reduced folates. As a way to increase the levels of tetrahydrobiopterin, in pregnant women with high blood pressure, women participating in the trial will take either a low dose or a high dose of a biologically-active form of reduced folate (tetrahydrofolate supplement) until delivery of their baby. A further group of women with high blood pressure will be recruited and will take a placebo. Blood tests will be taken and measurements performed to evaluate the heart and blood vessels of the participating women and their babies upon entry into the study and again at the time of birth. The investigators will also collect the umbilical cord and placenta tissue samples once the baby has been born, so that the investigators can assess blood vessel cell function following tetrahydrofolate supplementation in laboratory studies. In addition to the groups of women with high blood pressure, the investigators will also invite a group of women with an uncomplicated pregnancy to take part, as a comparison group, these women will not receive any supplementation. The investigators aim to investigate how levels of factors in the folate pathway differ in pregnant women with high blood pressure and if this is reflected in functional changes in the heart and blood vessels of these women. The investigators also aim to study whether this tetrahydrofolate supplement can increase the levels of tetrahydrobiopterin and if this improves blood vessel function. If successful, the investigators hope that the results of this study will enable us to design and conduct a larger study in future in order to test whether taking this tetrahydrofolate supplement will stop or reverse the changes caused by high blood pressure in pregnancy.

ELIGIBILITY:
Inclusion Criteria (Preeclampsia individuals):

* Diagnosed with preeclampsia, as defined in Section 8.1, at <34 weeks' gestation within the last 48 hours and with no delivery planned within the next week
* Receiving antenatal care in the John Radcliffe Hospital
* Participant is willing and able to give informed consent for participation in the study
* Age >18 and ≤45 years

Exclusion Criteria (Preeclampsia individuals):

The participant may not enter the study if ANY of the following apply:

Maternal

* History of cardiac impairments including uncontrolled arrhythmia, unstable angina, decompensated congestive heart failure or valve disease
* History of preexisting chronic renal disease
* Contraindication to taking folate related supplements
* Folate supplementation in excess of 400mcg in the third trimester
* Low vitamin B12 levels (<148 pmol/L)
* Intake of either proton pump inhibitors or anti-epileptic drugs
* Organ dysfunction Fetal
* Any known trisomy
* Fetus with congenital heart defect
* Fetus at a high risk of heart disease
* Known infection of fetus
* Known severe anaemia

Inclusion Criteria (Normotensive individuals):

* Participant is willing and able to give informed consent for participation in the study
* Age >18 and ≤45 years
* Normotensive, blood pressures <140/90 throughout antenatal period
* Less than 2 moderate risk factors for hypertensive disease in pregnancy according to the NICE guideline for management of hypertension in pregnancy
* SFlt/PIGF ratio <35

Exclusion Criteria (Normotensive individuals):

The participant may not enter the study if ANY of the following apply:

Maternal

* Diagnosis of hypertensive disorder of pregnancy
* Use of beta blockers such as atenolol or equivalent
* History of cardiac impairments including uncontrolled arrhythmia, unstable angina, decompensated congestive heart failure or valve disease
* History of preexisting chronic renal disease Fetal
* Any known trisomy
* Fetus with congenital heart defect
* Fetus at a high risk of heart disease
* Known infection of fetus
* Known severe anaemia

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 128 (Estimated)
Dates: Start 2021-06-01 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
To assess the change of maternal circulating BH4 biomarkers levels at baseline to prior to delivery. | Baseline (gestation approx. 28- 34 weeks) and prior to delivery
  Levels of BH4, Dihydrobiopterin (BH2), tetrahydrofolate, dihydrofolate reductase (DHFR), GTP cyclohydrolase I (GTPCH) will be assessed.
To assess the change of maternal nitric oxide levels at baseline to prior to delivery. | Baseline (gestation approx. 28- 34 weeks) and prior to delivery
  Levels of nitric oxide will be assessed in maternal serum samples.
To assess the levels of BH4 biomarkers in umbilical cord blood. | At delivery
  Levels of BH4, Dihydrobiopterin (BH2), tetrahydrofolate, dihydrofolate reductase (DHFR), GTP cyclohydrolase I (GTPCH) will be assessed in cord blood serum.
To assess the levels of BH4 biomarkers in placenta. | At delivery
  Levels of BH4, Dihydrobiopterin (BH2), tetrahydrofolate, dihydrofolate reductase (DHFR), GTP cyclohydrolase I (GTPCH) will be assessed in placental tissues.
To assess the levels of nitric oxide levels in umbilical cord blood. | At delivery
  Levels of nitric oxide will be assessed in cord blood serum.
To assess the levels of nitric oxide levels in placenta. | At delivery
  Levels of nitric oxide will be assessed in placental tissues.

SECONDARY OUTCOMES:
To assess whether maternal BH4 biomarkers levels are correlated with changes in the offspring. | Maternal: at baseline (gestation approx. 28- 34 weeks) and prior to delivery Umbilical cord and placenta: immediately after delivery
  Levels of folates, BH4 BH2, tetrahydrofolate, DHFR, and GTPCH will be assessed
To assess whether BH4 biomarkers levels are correlated with improved angiogenesis profile of maternal blood-derived endothelial cell forming colonies (ECFCs). changes in in-vitro maternal and fetal vascular function. | At baseline (gestation approx. 28- 34 weeks) and prior to delivery
  Angiogenesis profile of ECFCs (tube length, diameter, total area and duration for regression) will be determined via in vitro tube formation assay.
To assess whether BH4 biomarkers levels are correlated with improved angiogenesis profile of human umbilical vein endothelial cells (HUVECs). | At delivery
  Angiogenesis profile of HUVECs (tube length, diameter, total area and duration for regression) will be determined via in vitro tube formation assay.
To assess whether BH4 biomarkers levels are correlated with circulating angiogenic molecules (soluble fms-like tyrosine kinase-1 and placental growth factor). | At baseline (gestation approx. 34 weeks) and prior to delivery.
  Measurement of sFlt-1 and PlGF will be measure in serum samples in the clinical biochemistry laboratory.
To assess whether BH4 biomarkers levels are correlated with in-vivo flow-mediated dilatation (FMD) changes. | At baseline (gestation approx. 34 weeks) and prior to delivery.
  Brachial artery FMD induced by reactive hyperemia to assess vascular endothelial function.
To assess whether BH4 biomarkers levels are correlated with peripheral blood pressure changes. | At baseline (gestation approx. 34 weeks) and prior to delivery.
  Flow mediated dilatation, peripheral blood pressure, left and right ventricular mass and volumes and cardiac diastolic function.
To assess whether tetrahydrofolate levels are associated with cardiac remodelling. | At baseline (gestation approx. 34 weeks) and prior to delivery.
  Echocardiography will be performed and left and right ventricular mass and volumes and cardiac diastolic function will be investigated.
To investigate the acceptability and feasibility of taking the supplementation during pregnancy via questionnaire. | After delivery
  All participants will also be asked to complete a questionnaire assessing the acceptability of 5-MTHF supplementation. This questionnaire can be completed at any point before discharge.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Leeson, FRCP, Principal Investigator — University of Oxford, John Radcliffe Hospital
Locations (2):
- United Kingdom (2):
  - Oxford University Hospitals NHS Foundation Trust, Oxford, Oxfordhsire
  - Cardiovascular Clinical Research Facility, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Cutler HR, Kitt J, Sattwika PD, Finnigan LEM, Estevez-Fernandez A, Kenworthy Y, Suriano K, Frost A, Krasner S, Johnson C, McCourt A, Mills R, Tucker K, Cairns A, Roman C, Aye C, Mackillop L, Thilaganathan B, Chappell LC, Raman B, Lewandowski AJ, Lapidaire W, Leeson P. Subclinical Postpartum Renal Structure After Hypertensive Pregnancy Disorders. Hypertension. 2025 Nov;82(11):1948-1958. doi: 10.1161/HYPERTENSIONAHA.125.25130. Epub 2025 Aug 31. PMID 40886083
- See also: CAREFOL-HT Study — http://rdm.ox.ac.uk/carefol_ht